CLINICAL TRIAL: NCT04524065
Title: Effectiveness and Safety of an Early Mobilization Protocol in a Pediatric Intensive Care Unit
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Jeong Yi Kwon, Professor, Samsung Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 2020-05-136
Record Dates: First submitted 2020-08-19; First posted 2020-08-24 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: Critical Illness
Keywords: PICU; acute rehabilitation; early mobilization
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Early intervention group (Experimental): The 14 early rehabilitation sessions(10 physical therapy sessions; 15minutes per session, 4 occupational therapy sessions; 20minutes per session) occurred per week until discharge.
  Interventions: Other: Early rehabilitation protocol for children hospitalized in the PICU
- Control group (No Intervention): The control group received 2 sessions(physical therapy) per week over a 2-week period for 10 minutes each.

INTERVENTIONS:
Other: Early rehabilitation protocol for children hospitalized in the PICU — The early rehabilitation protocol was developed by a collaborative multidisciplinary team approach in Samsung Medical Center, and the central components include the involvement of physical therapy/occupational therapy (PT/OT).
  Arms: Early intervention group

SUMMARY:
This study evaluates the safety and effectiveness of an early rehabilitation program in a pediatric intensive care unit (PICU). Half of the participants will receive intensive and frequent an early mobilization program and others will receive conservative mobilization program.

DETAILED DESCRIPTION:
The 14 early rehabilitation sessions(10=physical therapy, 4=occupational therapy) occurred per week over a 2-week period (excluding weekends) in the early rehabilitation group for 15 minutes each. The control group received 2 sessions(physical therapy) per week over a 2-week period for 10 minutes each.

ELIGIBILITY:
Inclusion Criteria:

* Children admitted to the PICU due to critical illness
* Children aged 1-18 years

Exclusion Criteria:

* Increased intracranial pressure(ICP)
* History of brain surgery
* Children with fracture
* Admitted to the participating PICU ≤ 3 days
* Children with suspected brain death

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 142 (Estimated)
Dates: Start 2020-10-27 (Actual); Primary Completion 2025-08-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Change From Baseline Functional Status Score (FSS) at Post Test(PICU discharge) | Evaluation is conducted at two time points. At baseline (T0), assessment is carried out for within 7 days after admission to the PICU. For T1, assessment occurs within 7 days after PICU discharge or, for patients unable to be discharged, at the 30-da
  Functional Status Scale (FSS) domains of functioning included mental status, sensory functioning, communication, motor functioning, feeding, and respiratory status, categorized from normal (score = 1) to very severe dysfunction (score = 5). FSS scores ranged from 6 to 30.

SECONDARY OUTCOMES:
The Pediatric Evaluation of Disability Inventory-Computer Adaptive Test(PEDI-CAT) | Evaluation is conducted at two time points. At baseline (T0), assessment is carried out for within 7 days after admission to the PICU. For T1, assessment occurs within 7 days after PICU discharge or, for patients unable to be discharged, at the 30-da
  The PEDI-CAT incorporates a computer-adaptive platform with 276 items based on parental or caregiver reporting, and has four domains that cover daily activities, mobility, social/cognitive function, and responsibility. The PEDI-CAT yields a single score scaled from 0 to 100 for both Mobility and Self-care, with higher scores indicating greater function.
Duration of mechanical ventilation (days) | Perioid between intubation and extubation of mechanical ventilation
  Defined as the number of days of mechanical ventilation through an endotracheal tube during the PICU admission.
PICU length of stay (days) | From PICU admission to discharge
  Defined as the number of days of PICU length of stay.
Hospital length of stay (days) | From Baseline to hospital discharge
  Defined as the number of days of Hospital length of stay.
Number of patients discharged from the hospital to a place other than home | At hospital discharge
  Number of patients discharged from the hospital to a place other than home (rehabilitation facility).
Safety index | Evaluation is conducted at two time points. At baseline (T0), assessment is carried out for within 7 days after admission to the PICU. For T1, assessment occurs within 7 days after PICU discharge or, for patients unable to be discharged, at the 30-da
  * Frequency of thrombus and pressure sores occurred during intervention period
  * Frequency of abnormal vital signs occurred during intervention period
  * Frequency of any adverse events associated with intervention
The Pediatric Risk of Mortality III (PRISM III) | At PICU admission
  The PRISM III score has 17 physiologic variables subdivided into 26 ranges. The variables most predictive of mortality were minimum systolic blood pressure, abnormal pupillary reflexes, and stupor/coma. Other risk factors, including two acute and two chronic diagnoses, and four additional risk factors, were used in the final predictors. The PRISM III score and the additional risk factors were applied to the first 24 hours of stay (PRISM III-24).
Change From post-test(PICU discharge) Pediatric Quality of Life Inventory version 4.0 (PedsQL 4.0) at follow-up test(2 months) | Evaluation is conducted at two time points. At baseline (T0), assessment is carried out for within 7 days after admission to the PICU. For T1, assessment occurs within 7 days after PICU discharge or, for patients unable to be discharged, at the 30-da
  The Pediatric Quality of Life Inventory or PedsQLTM is a series of assessment instruments designed to measure the health-related quality of life of children. The PedsQL 4.0 provides an opportunity for the assessment of both overall (generic) quality of life as well as disease-specific quality of life.
  The PedsQL 4.0 Generic Core Scales are appropriate for assessing health-related quality of life in both healthy and chronically ill children. The four scales making up this generic battery include Physical Functioning (8 items), Emotional Functioning (5 items), Social Functioning (5 items), and School Functioning (5 items).
  A 5-point response scale is utilized across child self-report and parent proxy-report (0 = never a problem; 1 = almost never a problem; 2 = sometimes a problem; 3 = often a problem; 4 =almost always a problem).
Change From baseline The State-Trait Anxiety Inventory (STAI) at follow-up test(2 months) | Evaluation is conducted at two time points. At baseline (T0), assessment is carried out for within 7 days after admission to the PICU. For T1, assessment occurs within 7 days after PICU discharge or, for patients unable to be discharged, at the 30-da
  The State-Trait Anxiety Inventory (STAI) is a psychological inventory based on a 4-point Likert scale and consists of 40 questions on a self-report basis. The STAI measures two types of anxiety - state anxiety, or anxiety about an event, and trait anxiety, or anxiety level as a personal characteristic. Higher scores are positively correlated with higher levels of anxiety. STAI-X consists of 20 items each for measuring state anxiety and trait anxiety. Each item is rated on a 4-point scale (1 = Not at all, 4 = Very much so), with scores ranging from 20 to 80.
Canadian Occupational Performance Measure (COPM) | Evaluation is conducted at two time points. At baseline (T0), assessment is carried out for within 7 days after admission to the PICU. For T1, assessment occurs within 7 days after PICU discharge or, for patients unable to be discharged, at the 30-da
  At baseline, the interviewer assisted the child and family to identify occupational performance problems in the areas of self-care, productivity or leisure. Once they had identified these problems, they were written positively as goals, which participants and their parents then prioritised by importance on a scale from 1 to 10 (10 indicating greater importance). Scores out of 10 for self-perceived performance and satisfaction were then obtained from parent. The scores were summed and averaged over the number of priorities identified to produce two overall scores out of 10 for each participant: one for performance and one for satisfaction. At post-treatment and follow-up, participants were blinded to their previous ratings in order to limit potential bias. A 2 point change in score on the COPM is considered to be clinically meaningful.
Muscle strength measures of elbow flexor and knee extensor obtained with a hand-held dynamometer(MicroFET2). | Evaluation is conducted at two time points. At baseline (T0), assessment is carried out for within 7 days after admission to the PICU. For T1, assessment occurs within 7 days after PICU discharge or, for patients unable to be discharged, at the 30-da
  Maximal isometric voluntary contraction will be measured with a MicroFET2 hand-held dynamometer (Hoggan Indiustries, Inc., West Jordan, UT, USA). Maximal isometric muscle strength from two different muscle groups (knee extensors and elbow flexors) will be measured. It will be performed twice for each motion, and the higher one is derived as the result. Higher values indicates higher strength.
Pediatric Sequential Organ Failure Assessment(pSOFA) | Evaluation is conducted at two time points. At baseline (T0), assessment is carried out for within 7 days after admission to the PICU. For T1, assessment occurs within 7 days after PICU discharge or, for patients unable to be discharged, at the 30-da
  The Pediatric Sequential Organ Failure Assessment (pSOFA) score is a simple and objective score that allows for calculation of both the number and the severity of organ dysfunction in six organ systems (respiratory, coagulatory, liver, cardiovascular, renal, and neurologic) and the score can measure individual or aggregate organ dysfunction. Daily pSOFA score is the sum of the 6 subscores and higher scores indicate a worse outcome. Score assesses 6 organ systems: respiratory, hematological, hepatic, cardiovascular, neurological and renal. A subscore of 0 (normal)-4(most abnormal) points.

CONTACTS AND LOCATIONS:
Overall Officials: Jeong-Yi Kwon, PhD, Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, South Korea